CLINICAL TRIAL: NCT06259903
Title: A Single Center, Single Dose, Double-blind, Randomized, Placebo-Controlled, Dose-Escalating Study to Evaluate Safety, Tolerability and Pharmacokinetics of Subcutaneously Administered MD-18 in Healthy Subjects.
Brief Title: Subcutaneous Administration of MD-18 in Healthy Subjects
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Cohen Global, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: MD-18-01
Record Dates: First submitted 2024-01-29; First posted 2024-02-14 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Intervention Model Description: Five subjects in cohort 1 will be administered a single subcutaneous dose of 40 mg MD-18 and two will receive placebo. The cohort will be staggered with 2 active and one placebo patient treated on day 1 and the remainder on Day 3 if there are no safety concerns. The same dosing regimen will be observed for each incremental cohort, with the remaining planned doses being 80, 160, 240 and 320 milligram (mg).
Who Masked: Participant, Investigator
Masking Description: Study medication will be supplied in labelled vials, clearly identifying the contents and indicating that the product is an investigational drug. An unblinded pharmacist at the clinical site will be responsible for drawing up the appropriate amount of study medication into a syringe and labelling the syringe for administration to the specific patient according to the randomization scheme.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- 40 milligram (mg) MD-18 OR 40 milligram(mg) Placebo (Experimental): A single dose of subcutaneous injection of 40mg MD-18 OR 40mg Placebo will be given on day zero.
  Interventions: Drug: MD-18
- 80 milligram (mg) MD-18 OR 80 milligram (mg) Placebo (Experimental): A single dose of subcutaneous injection of 80mg MD-18 OR 80mg Placebo will be given on day zero.
  Interventions: Drug: MD-18
- 160 milligram (mg) MD-18 OR 160 milligram (mg) Placebo (Experimental): A single dose of subcutaneous injection of 160mg MD-18 OR 160mg Placebo will be given on day zero.
  Interventions: Drug: MD-18
- 240 milligram (mg) MD-18 OR 240 milligram (mg) Placebo (Experimental): A single dose of subcutaneous injection of 240mg MD-18 OR 240mg Placebo will be given on day zero.
  Interventions: Drug: MD-18
- 320 milligram (mg)MD-18 OR 320 milligram (mg) Placebo (Experimental): A single dose of subcutaneous injection of 320mg MD-18 OR 320mg Placebo will be given on day zero.
  Interventions: Drug: MD-18

INTERVENTIONS:
Drug: MD-18 — Subcutaneous Administration of MD-18 in Healthy Subjects.

SUMMARY:
A Single Center, Single Dose, Double-blind, Randomized, Placebo-controlled Dose-Escalating Study to Evaluate Safety, Tolerability and Pharmacokinetics of Subcutaneously Administered MD-18 in healthy subjects.

DETAILED DESCRIPTION:
This study will be conducted as a single-center study. A single escalating dose of MD-18 will be administered to each subject with a seven-day follow-up. 35 subjects will be enrolled. Cohorts will receive doses of 40. 80, 160, 240 or 320 milligram of MD-18 using 5:2 (active: placebo) randomization. Sentinel dosing will be used, consisting of enrolling three subjects at a 2:1 active to placebo ratio followed by the remaining subjects in the respective dose cohorts enrolled 48 hours later. Each of the 5 dose cohorts will enroll five active and two placebo subjects, with a total of 25 subjects receiving active therapy across the 5 arms and 10 subjects receiving placebo. The study will be conducted on an in-patient basis for the first 24 hours, followed by discharge and telephone check-in at 48 and 72 hours and return for follow-up visit at 7 days after administration of a single dose of MD-18.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 18-70 years, both genders.
2. Healthy as determined by a physician, based on history, medical examination, vital signs, laboratory tests, cardiac monitoring and respiratory function. History must comply with the following:

   1. Absence of clinically significant illness or surgery within the preceding 12 weeks.
   2. Absence of clinically significant history of neurological, endocrine, cardiovascular, pulmonary, hematological, immunologic, psychiatric, gastrointestinal, renal, hepatic, and/or metabolic disease.
3. Male subjects with female partners of childbearing potential must agree to utilize an approved contraceptive during the study.
4. Female subjects of child-bearing potential with negative urine pregnancy tests and who agree to use contraception during the study.
5. Female subjects of non-child-bearing potential (i.e. tubal ligation, hysterectomy, or postmenopausal).
6. Body mass index (BMI) of 18.5-39.9 kg/m2

Exclusion Criteria:

1. History of excessive alcohol use (defined as >21 drinks per week for males and >14 drinks per week for females), recreational drug use or drugs of abuse within the past three months, or failure on urinary drug screen. Note: use of Cannabinoids for medical purposes is allowed.
2. Pregnant or breastfeeding within six months of screening assessment.
3. Substantial changes in eating habits or exercise routine within the preceding three months.
4. Evidence of eating disorders.
5. >5% weight change in the past three months.
6. Bariatric surgery within the past five years.
7. Significant renal impairment glomerular filtration rate (GFR) <60 milligram/milliliter/1.73m2).
8. Liver function tests (i.e., alanine aminotransferase, Aspartate Amino Transferase, alkaline phosphatase) greater than twice the upper limit of normal upon repeated measurements.
9. Diseases interfering with metabolism and/or ingestive behavior (e.g., myxedema, Cushing's disease, schizophrenia, major psychoses, unmanaged depression).
10. Use of drugs approved for the treatment of obesity.
11. Any clinically significant abnormality following the Investigator's review of the physical examination and clinical laboratory tests.
12. A baseline prolongation of ventricular activation and recovery interval after repeated measurements of >450 millisecond; a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS).
13. Participation in an investigational drug trial within three months prior to dosing in the present study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by the collection of Adverse Events. | For all study duration (approximately two months).
  Adverse Events Collection.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by the collection of pre and post dose pharmacokinetics samples. | Before and after dose administration on Days 0 and 1.
  Pharmacokinetics sampling is predicated on a T1/2 less than 6 hours to enable inpatient monitoring for 4-5 half-lives.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by the collection of vital signs. | On screening visit and on days 1 and 7.
  Systolic and diastolic blood pressure in millimeters of mercury, Heart rate in beats per minute, Respiratory rate in breath per minute.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by the collection of Lab samples. | On screening visit and on days 1 and 7.
  Collection of Complete blood count, Serum chemistry, Coagulation panel and Urine analysis.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by the collection of anthropometric measurement's. | On screening visit and on days 1 and 7. (height will be collected only in the screening visit).
  Weight in kilograms, Height in meters.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by an electrocardiogram examination. | On screening visit and on days 0,1 and 7.
  12-lead ECG will be obtained within 1 hour before and 3 hours (+15 minutes) after dosing and prior to discharge. The ECG machine will automatically calculate the heart rate, measure of the time from the beginning of the atrial depolarization to the beginning of the ventricular depolarization, depolarization of ventricles and time taken for ventricular depolarization and repolarization. At each time-point, ECG will be obtained in triplicate.
To determine the safety of a single subcutaneously administered dose of MD-18 in healthy subjects, as assessed by physical examination. | On screening visit and on days 1 and 7.
  A complete physical examination (head, eyes, ears, nose and throat, heart, lungs, abdomen, skin, cervical and axillary lymph nodes, neurological, and musculoskeletal systems) will be performed.

SECONDARY OUTCOMES:
Analysis of pharmacokinetics samples of MD-18 by lab methods. | Before and after dose administration on Days 0 and 1.
  A pharmacokinetics analysis will be conducted if plasma concentrations exceed the lower limit of quantitation of 5 nanogram/milliliter using a validated and a model-independent methods.

OTHER OUTCOMES:
Treatment-emergent Adverse Events (TEAEs) will be assessed. | For all study duration ( approximately two months).
  Number of Participants with Treatment-emergent Adverse Events (TEAEs) as assessed by the CTCAE v5.0.
Tolerability (referred to as the dose-limiting tolerability) will be assessed by the number of reported cases with nausea and injection site reaction. | On days 0-3.
  Will be assessed by the number of reported cases with nausea and injection site reaction according to the following time frames:
  1. Severe nausea within 24 hours of taking drug
  2. Severe injection site reaction within 72 hours (grade ≥3)
Adverse events of special interest will be assessed. | For all study duration ( approximately two months).
  Assessment of the frequency of clinical symptoms of nausea, vomiting, and injection site discomfort or irritation.

CONTACTS AND LOCATIONS:
Overall Officials: Amir Tirosh, Prof, Study Chair — Cohen Global, Ltd.
Locations (1):
- Sheba Medical Center, Ramat Gan, Please Select, Israel

IPD SHARING:
Plan to Share IPD: No